CLINICAL TRIAL: NCT07263347
Title: Prospective Observational Study of Perioperative Biomarkers and Outcomes in Deep Inferior Epigastric Perforator (DIEP) Flap Breast Reconstruction
Brief Title: DIEP Flap Breast Reconstruction: Perioperative Biomarkers and Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xinhong Wu, PhD, vice-president, Hubei Cancer Hospital
Other Study IDs: LLHBCH2025YN-075
Record Dates: First submitted 2025-09-27; First posted 2025-12-04 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasms; Ischemia-Reperfusion Injury; Postoperative Complications; Wound Healing; Oxidative Stress; Inflammation
Keywords: Deep inferior epigastric perforator (DIEP) flap; Autologous breast reconstruction; Free tissue transfer; Ischemia-reperfusion injury
MeSH Terms: conditions — Breast Neoplasms; Reperfusion Injury; Postoperative Complications; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Only acellular fractions from DIEP patients' peripheral blood will be retained: serum (clot-activator tube) and EDTA plasma supernatant. Samples will be centrifuged to remove cells and platelets (platelet-poor plasma as needed), aliquoted, and stored at -80°C for inflammation/oxidative-stress protein and metabolite assays (e.g., IL-6, TNF-α, IL-10, MDA, SOD, CAT, VEGF, D-dimer, lactate, LDH). No long-term retention of whole blood, buffy coat/nucleated cells, PBMCs, saliva, urine, tissue, or swabs; any leftover whole blood from clinical labs will be destroyed per policy. All human specimens are de-identified and labeled with study IDs. No DNA/RNA extraction or sequencing will be performed on any retained human specimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DIEP flap reconstruction patients (longitudinal peripheral blood cohort): Prospective observational cohort of women (18-70 years) undergoing immediate autologous breast reconstruction with a DIEP free flap. Standard peri-operative care only; no investigational imaging or drug (no Mn/QD-SAC) is administered. Serial peripheral blood is collected at pre-op baseline (≤24 h) and at 0 h, 6 h, 24 h, and 72 h post-op (≈10 mL/timepoint; serum + EDTA plasma). Primary measurement is plasma IL-6; additional analytes include IL-1β, TNF-α, IL-8, IL-10, IL-18, HMGB1, vWF, VEGF, HIF-1α, MDA, 8-iso-PGF2α, SOD, CAT, GSH-Px, lactate, LDH, PT/APTT/fibrinogen, D-dimer, and CBC. Samples are processed within 2 h and stored at -80°C for batch ELISA/biochemical assays. Clinical data (age, BMI, operative/ischemia times, flap perfusion assessments, complications, fat necrosis/partial flap loss) are recorded. Target enrollment ~30 participants.

SUMMARY:
Brief Summary This observational study will follow patients who undergo DIEP flap breast reconstruction to better understand a common surgical challenge called ischemia-reperfusion (I/R) injury. I/R injury can happen when a flap has a period without blood flow (ischemia) and then blood flow returns (reperfusion). This process may trigger inflammation and oxidative stress and is associated with fat necrosis or partial flap loss.

1. What is being studied

1. The investigators will measure inflammation and oxidative stress markers in blood (for example, interleukin-6 [IL-6]) from before surgery through the first 72 hours after surgery.
2. These data will help map the normal and abnormal patterns of recovery after surgery and may inform future approaches to monitoring and protecting flap tissue.
3. No experimental drug or device is given to participants in this study. Separate animal studies are developing a near-infrared imaging and antioxidant nanomaterial (Mn/QD-SAC); this is not used in participants here.

2. Who can take part

1. Women aged 18-70 scheduled for immediate DIEP flap breast reconstruction after breast cancer surgery.
2. Key exclusions include severe heart, liver, or kidney disease; significant clotting problems; active infection or autoimmune disease; long-term use of immunosuppressants/anti-inflammatory drugs; pregnancy or breastfeeding; or other reasons judged by the research team.

3. What will happen if you join

1. After providing informed consent, participants will have blood drawn at five time points: pre-operative baseline (within 24 hours before surgery) and at 0, 6, 24, and 72 hours after surgery (about 10 mL each time; total ~50 mL).
2. Blood will be processed and stored under secure conditions and tested for inflammation and oxidative stress markers.
3. The investigators will also record routine clinical information from the medical record (such as age, BMI, surgery duration, ischemia time, and clinical assessments of flap outcomes and complications).
4. Participation does not change the participant's clinical care before, during, or after surgery.

4. Risks and benefits

1. Risks are those of standard blood draws: brief pain, bruising, bleeding, dizziness, and rare infection.
2. There is no direct medical benefit to participants. Results may help improve understanding and future care for patients undergoing flap reconstruction.

5. Privacy and data protection

1. Samples and data will be coded without names. Identifying information is stored separately with restricted access.
2. Research results are not routinely added to the medical record or returned to participants unless a finding has clear, actionable clinical significance and is approved by the ethics committee.

6. Time commitment and costs

1. All blood draws occur during the routine hospital stay. There is no additional follow-up required after discharge.
2. There is no cost to participate.

7. Voluntary participation Joining the study is voluntary. Participants may withdraw at any time without affecting their medical care.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 18-70 years old.
2. Clinically diagnosed with breast cancer and scheduled for immediate DIEP free-flap breast reconstruction after mastectomy.
3. Conscious and able to understand and voluntarily sign written informed consent.

Exclusion Criteria:

1. Severe cardiac, hepatic, or renal dysfunction or severe coagulopathy (e.g., NYHA class III-IV, Child-Pugh class C, eGFR <30 mL/min/1.73 m²).
2. Preoperative active infection, autoimmune disease, or long-term use of immunosuppressants/anti-inflammatory drugs (e.g., corticosteroids).
3. Pregnant or breastfeeding.
4. Prior ipsilateral breast surgery or radiotherapy that may affect local blood circulation assessment.
5. Any condition deemed unsuitable by the investigator (e.g., poor compliance).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adult women (18-70 years) with breast cancer at Hubei Cancer Hospital undergoing mastectomy with immediate DIEP free-flap breast reconstruction. Approximately 30 consecutive eligible patients able to provide written informed consent will be enrolled. Exclusions include severe cardiac/hepatic/renal dysfunction or severe coagulopathy, preoperative active infection, autoimmune disease or chronic immunosuppressive/anti-inflammatory therapy (e.g., corticosteroids), pregnancy or breastfeeding, and prior ipsilateral breast surgery or radiotherapy. This is an observational perioperative biomarker cohort; no investigational agents or devices are administered.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Viable DIEP flap area (%) at postoperative day 7 | Postoperative day 7
  Standardized digital photographs will be obtained on POD7 under uniform lighting and distance with a calibration ruler. Viable flap area (%) is calculated as [viable area/total area]×100 using blinded planimetry by two independent raters; discrepancies >5% are adjudicated by a third rater. This endpoint reflects clinical benefit and flap survival. This is a co-primary endpoint with IL-6; the family-wise error rate is controlled at 0.05 using the Bonferroni correction (two-sided α=0.025 per endpoint).
Plasma interleukin-6 (IL-6) concentration at 24 hours after surgery | Baseline (up to 24 hours before surgery) and 24 hours after surgery.
  Plasma IL-6 (pg/mL) will be quantified in EDTA plasma using a validated sandwich enzyme-linked immunosorbent assay (ELISA). Blood is drawn up to 24 hours prior to surgery (baseline) and at 24 hours after surgery; plasma is separated within 2 hours, aliquoted, and stored at -80°C (single freeze-thaw). Samples are run in duplicate with a 7-point standard curve and quality control samples. The co-primary analysis will focus on the change in IL-6 from baseline to 24 hours post-surgery, analyzed as a continuous variable with prespecified covariates (age, body mass index, ischemia time, operative duration). This endpoint is co-primary with flap viability; the Bonferroni-adjusted family-wise error rate is 0.05 (two-sided alpha=0.025).

SECONDARY OUTCOMES:
Plasma tumor necrosis factor alpha (TNF-α) concentration at 24 hours after surgery | Baseline (up to 24 hours before surgery) and 24 hours after surgery.
  EDTA plasma TNF-α (pg/mL) will be quantified using a validated sandwich ELISA. Blood is drawn up to 24 hours prior to surgery (baseline) and at 24 hours after surgery; plasma is processed within 2 hours, aliquoted, and stored at -80°C (single freeze-thaw). Samples are run in duplicate. The primary analysis will assess the change in TNF-α from baseline to 24 hours post-surgery as a continuous variable.
Plasma interleukin-10 (IL-10) concentration at 24 hours after surgery | Baseline (up to 24 hours before surgery) and 24 hours after surgery.
  EDTA plasma IL-10 (pg/mL) will be quantified using a validated sandwich ELISA. Blood is drawn up to 24 hours prior to surgery (baseline) and at 24 hours after surgery; plasma is separated within 2 hours, aliquoted, and stored at -80°C (single freeze-thaw). Samples are run in duplicate. The analysis will focus on the change in IL-10 concentration from baseline to 24 hours post-surgery as a continuous variable.
Area under the curve (AUC) for plasma malondialdehyde from baseline to 24 hours after surgery | Baseline (up to 24 hours before surgery), 6 hours after surgery, and 24 hours after surgery.
  Plasma malondialdehyde will be measured using a validated thiobarbituric acid reactive substances assay. Blood is collected up to 24 hours prior to surgery (baseline), and at 6 hours and 24 hours after surgery; plasma is processed within 2 hours, aliquoted, and stored at -80°C (single freeze-thaw). The area under the concentration-time curve from baseline to 24 hours after surgery will be calculated using the linear trapezoidal method based on the values at the three time points, and analyzed as a continuous variable.
Area under the curve (AUC) for plasma superoxide dismutase activity from baseline to 24 hours after surgery | Baseline (up to 24 hours before surgery), 6 hours after surgery, and 24 hours after surgery.
  Superoxide dismutase activity will be measured using a validated enzymatic activity kit. Blood collection and processing as per Outcome 5. The AUC from baseline to 24 hours will be calculated and analyzed separately as a continuous variable.
Area under the curve (AUC) for plasma glutathione peroxidase activity from baseline to 24 hours after surgery | Baseline (up to 24 hours before surgery), 6 hours after surgery, and 24 hours after surgery.
  Glutathione peroxidase activity will be measured using a validated enzymatic activity kit. Blood collection and processing as per Outcome 5. The AUC from baseline to 24 hours will be calculated and analyzed separately as a continuous variable.
Number of participants with surgical site infection within 30 days | From surgery to postoperative day 30
  Infection at the flap or donor site meeting CDC criteria (e.g., purulent drainage, positive culture, or surgeon diagnosis requiring treatment). Data will be captured prospectively from medical records and follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to patient privacy and ethical considerations, absence of consent for data sharing, institutional/regulatory restrictions, and limited resources for secure de-identification and data hosting. Aggregate results will be available in publications or upon request.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT07263347/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT07263347/ICF_001.pdf